CLINICAL TRIAL: NCT02114203
Title: A Phase 1b, Randomized, Double-blind (Sponsor Open), Placebo Controlled Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Pf 04447943, Co-administered With And Without Hydroxyurea, In Subjects With Stable Sickle Cell Disease
Brief Title: Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Study Of PF-04447943, Co-Administered With And Without Hydroxyurea, In Subjects With Stable Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Basic Science
Other Study IDs: B0401016; 2014-001677-13 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-07

CONDITIONS: Phase 1 Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- cohort 1 PF-04447943 (Experimental)
  Interventions: Drug: PDE9i
- cohort 2 PF-04447943 (Experimental)
  Interventions: Drug: PDE9i
- placebo comparator (Placebo Comparator)
  Interventions: Drug: placebo for PDE9i
- optional cohort of PF-04447943 (Experimental)
  Interventions: Drug: PDE9i

INTERVENTIONS:
Drug: PDE9i — oral dose, every 12 hours for 28 days
  Arms: cohort 1 PF-04447943; optional cohort of PF-04447943
Drug: PDE9i — oral dose, every 12 hours for 28 days
  Arms: cohort 2 PF-04447943; optional cohort of PF-04447943
Drug: placebo for PDE9i — oral dose, every 12 hours for 28 days
  Arms: placebo comparator
Drug: PDE9i — oral dose, every 12 hours for 28 days
  Arms: optional cohort of PF-04447943

SUMMARY:
This study is being conducted to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of an investigational drug, PF-04447943, in subjects with stable sickle cell disease with and without co-administration with hydroxyurea. This study will also aid in selecting the doses for future studies and evaluation of substances in the blood which may help access the effectiveness of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with a confirmed diagnosis of sickle cell disease (HbSS or HBS-β0 thalassemia) between the ages of 18 and 65 years, inclusive
* Subjects who are being treated with hydroxyurea must be on a stable dose for at least 8 weeks, with the intent of remaining on the same dose of hydroxyurea throughout the clinical trial including the protocol-specified follow-up period. Subjects who are not treated with hydroxyurea should not plan to begin treatment during the study period.
* Body Mass Index (BMI) of 17.5 to 35 kg/m2; and a total body weight >40 kg (88 lbs

Exclusion Criteria:

* History of a recent major surgery, within 3 months of baseline visit.
* Serious infection (requiring hospitalization or parenteral antibiotics) within 1 month of baseline visit.
* History of cerebrovascular accident or seizure disorder.
* Subjects with a history of clinically significant orthostatic blood pressure (BP) changes or clinically significant orthostatic symptoms.
* Known previous diagnosis of acute hepatitis of any aetiology Hepatitis B or C or Human immunodeficiency virus (HIV) infection.
* History of any malignancy except for subjects who had a basal or squamous cell cancer which has been treated and fully resolved for a minimum of 5 years.
* History or evidence of cardiac disease including: myocardial infarction, cardiac arrhythmia
* Systemic therapy with any of the following medications that are strong or moderate CYP3A4 inhibitors within 7 days or 5 half-lives (whichever is longer) or CYP3A inducers within 28 days prior to the first dose of the trial medication, or during the trial.
* Use of PDE5 inhibitors within 7 days prior to the first dose of the trial medication, or at any time during the trial.
* Creatinine clearance <30ml/min.
* Hemoglobin level <6 gm/dL.
* Alanine transaminase (ALT/SGPT) and Aspartate aminotransferase (AST/SGOT) >2x upper limit of normal, (based on clinic laboratory normal range).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen for illicit drug.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 2 months (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 or a QRS interval >120 msec msec at Screening.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* A family history of long QT syndrome and/or ECG abnormalities at screening or randomization, including those listed below:

  * Subjects with pre-randomization evidence of QTcF prolongation (defined as >450 ms) at screening or baseline are not eligible for randomization.
  * Predominant heart rhythm other than normal sinus rhythm eg, atrial fibrillation, atrial flutter, supraventricular tachycardia.
  * Atrioventricular (AV) block greater than first degree.
* Use of concomitant medications that prolong the QT/QTc interval
* Pregnant females and, breast feeding females and females of childbearing potential; male and female subjects of childbearing potential who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 30 days after the last dose of investigational product.
* Subjects who lack the capacity to consent for themselves.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (10):
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - Boston Medical Center E7E, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Interfaith Medical Center, Brooklyn, New York
  - UNC Hospitals' Investigational Drug Service Pharmacy, Chapel Hill, North Carolina
  - UNC School of Medicine Clinical and Translational Research Center, Chapel Hill, North Carolina
  - Investigational Drug Services, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Pfizer Clinical Research Unit, Brussels, Belgium
- Italy (2):
  - Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - A.O.O.R Villa Sofia - V. Cervello, Palermo
- Centre for Human Drug Research, Leiden, Netherlands
- United Kingdom (7):
  - Royal Liverpool and Broadgreen University Hospital Trust, Liverpool, Merseyside
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Manchester Royal Infirmary, Manchester
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- [Derived] Charnigo RJ, Beidler D, Rybin D, Pittman DD, Tan B, Howard J, Michelson AD, Frelinger AL , III, Clarke N. PF-04447943, a Phosphodiesterase 9A Inhibitor, in Stable Sickle Cell Disease Patients: A Phase Ib Randomized, Placebo-Controlled Study. Clin Transl Sci. 2019 Mar;12(2):180-188. doi: 10.1111/cts.12604. Epub 2018 Dec 31. PMID 30597771
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401016&StudyName=Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Study%20Of%20PF-04447943%2C%20Co-Administered%20With%20And%20Without%20Hydroxyurea%2C%20In%20Subj

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, a total of 30 potential participants were randomized to the study, and 29 of them were assigned to and received study treatment, 1 participant in the PF-04447943 25 mg twice daily (BID) treatment group withdrew from the study after randomization but prior to study treatment.
Groups:
- PF-04447943 5 mg BID: PF-04447943 tablet was administered orally at 5 mg twice daily (BID) for up to 29 days.
- PF-04447943 25 mg BID: PF-04447943 tablet was administered orally at 25 mg twice daily (BID) for up to 29 days.
- Placebo: Placebo matched to PF-04447943 tablet was administered orally twice daily (BID) for up to 29 days.
Period: Overall Study
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Started | 7 | 16 | 7
Completed | 7 | 14 | 7
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo | Total
Number analyzed (Participants) | 7 | 16 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (10.6) | 36.3 (11.0) | 39.4 (14.0) | 37.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 5 | 18
  Male | 4 | 6 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Change From Baseline in Vital Signs
Description: Number of participants with changes from baseline in vital signs meeting the following criteria is presented: (1) maximum increase from baseline in supine systolic blood pressure (SBP) >=30 millimeters of mercury (mmHg); (2) maximum increase from baseline in supine diastolic blood pressure (DBP) >=20 mmHg; (3) maximum decrease from baseline in supine SBP >=30 mmHg; and (4) maximum decrease from baseline in supine DBP >=20 mmHg.
Time Frame: Baseline up to 30 days post last dose on Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants
  Maximum increase in supine SBP >=30 mmHg | 0 | 0 | 0
  Maximum increase in supine DBP >=20 mmHg | 2 | 0 | 1
  Maximum decrease in supine SBP >=30 mmHg | 0 | 1 | 0
  Maximum decrease in supine DBP >=20 mmHg | 2 | 0 | 1

2. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Change From Baseline in Neurologic Function
Description: Clinical assessment of neurologic functions included cranial nerve function, coordination, deep tendon reflexes, muscle strength, and reflexes (left and right ankles). Clinical importance of neurologic function changes was determined by the investigator.
Time Frame: Baseline up to Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Change in Physical Examination Findings
Description: Physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Clinical importance of physical examination changes was determined by the investigator.
Time Frame: Baseline up to 30 days post last dose on Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Treatment-Emergent Electrocardiogram (ECG) Findings
Description: Maximum absolute values and increases from baseline were summarized for PR interval (time from the beginning of P wave to the start of QRS complex, corresponding to the end of atrial depolarization and onset of ventricular depolarization), QRS complex (time from Q wave to the end of S wave, corresponding to ventricle depolarization), and QTcF interval (time from the beginning of Q wave to the end of T wave corresponding to electrical systole corrected for heart rate using Fridericia's formula). Number of participants with ECG findings meeting the following criteria is presented: (1) PR interval >=300 msec; (2) QRS complex >=200 msec; (3) QTcF interval: 450 to <480 msec; (4) QTcF interval: 480 to <500 msec; (5) QTcF interval >=500 msec; (6) PR interval percent increase from baseline >=25/50 percent; (7) QRS complex percent increase from baseline >=25/50 percent; (8) QTcF interval increase from baseline: 30 to <60 msec; (9) QTcF interval increase from baseline >=60 msec.
Time Frame: Baseline up to 30 days post last dose on Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants
  Maximum PR interval >=300 msec | 0 | 0 | 0
  Maximum QRS complex >=200 msec | 0 | 0 | 0
  Maximum QTcF interval: 450 to <480 msec | 0 | 3 | 2
  Maximum QTcF interval: 480 to <500 msec | 0 | 0 | 1
  Maximum QTcF interval: >=500 msec | 0 | 0 | 0
  PR interval increase >=25/50 percent | 0 | 0 | 0
  QRS complex increase >=25/50 percent | 0 | 0 | 0
  QTcF interval increase: 30 to <60 msec | 0 | 1 | 0
  QTcF interval increase >=60 msec | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Change From Baseline in Symptoms of Sickle Cell Disease
Description: The following symptoms were assessed: anemia; fatigue; chronic pain; acute pain; infections; fever; swelling hands; swelling feet; abdominal swelling; pale skin; pale nail beds; yellow tint to skin; whites of eyes turned yellow; stroke. Number of participants with changes from baseline deemed potentially clinically important by the investigator is presented.
Time Frame: Baseline up to 30 days post last dose on Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of its causal relationship with study treatment. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; was life-threatening (immediate risk of death); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study drug and up to follow-up visit (30 days post last dose on Day 29) that were absent before treatment or that worsened after treatment. AEs included both serious and non-serious AEs.
Time Frame: Day 1 to 30 days post last dose on Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants
  AEs | 7 | 13 | 7
  SAEs | 2 | 1 | 0
  Withdrawal due to TEAEs | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: The laboratory test included: hematology (hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet count, white blood cell count, absolute total neutrophils, eosinophils, monocytes, basophils, and lymphocytes), chemistry (blood urea nitrogen/urea, serum creatinine, fasting glucose, calcium, sodium, potassium, chloride, total carbon dioxide, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, and high sensitivity C-reactive protein), urinalysis (pH, qualitative glucose, qualitative protein, qualitative blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, and microscopy), and other tests (follicle stimulating hormone and serum human chorionic gonadotropin, urine drug screening). Abnormality was determined by the investigator.
Time Frame: Baseline up to 30 days post last dose on Day 29
Population: The safety analysis population was defined as all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Number analyzed (Participants) | 7 | 15 | 7
participants | 7 | 15 | 7

8. Secondary Outcome: Area Under the Curve From Time Zero to 12 Hours Post Dose (AUC(0-12h)) of PF-04447943
Description: AUC(0-12h) referred to area under the plasma concentration-time curve from 0 to 12 hours post dose.
Time Frame: Prior to 0 hour, and 0.5, 1, 2, 4, 8, and 12 hours post dose on Day 1
Population: The full analysis set (FAS) was used for all PK analyses, and it included all participants randomized to treatment who had taken at least 1 dose of study medication. Data for this outcome measure were not planned to be analyzed for the placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID
Number analyzed (Participants) | 7 | 15
nanogram*hour/milliliter | 242.0 (35) | 1170 (29)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04447943
Time Frame: Prior to 0 hour, and 0.5, 1, 2, 4, 8, and 12 hours post dose on Day 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID
Number analyzed (Participants) | 7 | 15
ng/mL | 45.83 (39) | 248.2 (31)

10. Secondary Outcome: Time for Maximum Observed Plasma Concentration (Tmax) of PF-04447943
Time Frame: Prior to 0 hour, and 0.5, 1, 2, 4, 8, and 12 hours post dose on Day 1
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID
Number analyzed (Participants) | 7 | 15
hours | 1.92 [1.00 to 4.00] | 1.00 [0.500 to 4.05]

ADVERSE EVENTS:
Time Frame: Day 1 to follow-up visit (30 days post last dose on Day 29)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-04447943 5 mg BID | PF-04447943 25 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/15 | 0/7
Other Adverse Events (participants affected / at risk) | 7/7 | 13/15 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04447943 5 mg BID (N=7) | PF-04447943 25 mg BID (N=15) | Placebo (N=7)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04447943 5 mg BID (N=7) | PF-04447943 25 mg BID (N=15) | Placebo (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1 | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 2 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 6 | 2
Gait disturbance (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Tenderness (General disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood pressure systolic increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 4 | 5 | 2
Lethargy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.